CLINICAL TRIAL: NCT05222620
Title: Phase IIR Trial of Single Fraction Stereotactic Radiosurgery (SRS) Compared With Fractionated SRS (FSRS) for Intact Metastatic Brain Disease (FRACTIONATE)
Brief Title: SRS Compared With FSRS for Treatment of Intact Metastatic Brain Disease, FRACTIONATE Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2163; NCI-2021-14230 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-003768 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-01-11; First posted 2022-02-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (single fraction SRS) (Other): Patients undergo single fraction SRS.
  Interventions: Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery; Procedure: Magnetic Resonance Imaging
- Arm B (fractionated SRS) (Other): Patients undergo fractionated SRS.
  Interventions: Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo single fraction SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery; SRS
  Arms: Arm A (single fraction SRS)
Radiation: Stereotactic Radiosurgery — Undergo fractionated SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery; SRS
  Arms: Arm B (fractionated SRS)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MRI; MR Imaging; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial compares the effect of single fraction stereotactic radiosurgery to fractionated stereotactic radiosurgery for the treatment of patients with cancer that has spread to the brain (metastatic brain disease). Stereotactic radiosurgery (SRS) is a form of radiation therapy that focuses high-power energy on a small area of the body. This trial is being done to determine if single (one) fraction stereotactic radiosurgery is better than fractionated stereotactic radiosurgery or vice versa in controlling tumor and side effects in patients with tumors that have spread to the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To ascertain if the composite endpoint of cumulative treatment failure, defined by time to either local failure or symptomatic radiation brain necrosis of the largest brain metastasis (target lesion), is increased with fractionated stereotactic radiosurgery (FSRS) compared to single fraction stereotactic radiosurgery (SSRS).

SECONDARY OBJECTIVES:

I. To ascertain whether there is improved overall survival in patients who undergo FSRS compared to patients who receive SSRS.

II. To tabulate and descriptively compare the post-treatment adverse events associated with the interventions, including the potential impact of immunotherapy and targeted therapy.

III. To compare rates of radiation necrosis in patients who receive FSRS to patients who receive SSRS.

IV. To evaluate if there is any difference in central nervous system (CNS) failure patterns (e.g. local, distant brain failure) in patients who receive FSRS compared to patients who receive SSRS.

V. To ascertain whether FSRS prolongs time to neurologic death as compared to SRS.

VI. To determine whether there is improved patient reported outcomes (Functional Assessment of Cancer Therapy [FACT]-Brain Symptom Index [FBrSI]-24) including quality of life for patients who receive FSRS compared to patients who receive SSRS.

VII. To evaluate if there is any difference in CNS failure patterns (e.g. local, distant brain failure) and symptomatic radiation necrosis rates in patients who are treated with gamma knife compared to patients who are treated with a linear accelerator platform.

VIII. To determine whether differences in time to local failure, time to necrosis, or their composite endpoint cumulative treatment failure differs between treatment arms (or other patient or treatment factors) when analyzed on a "per lesion" basis rather than the per patient basis utilized for the primary endpoint.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo single fraction SRS. Patients also undergo magnetic resonance imaging (MRI) at screening and during follow up.

ARM B: Patients undergo fractionated SRS. Patients also undergo MRI at screening and during follow up.

After completion of study treatment, patients are followed up at 3 months, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Presence of presumed brain metastases from an extra-cerebral tumor site (e.g. lung, breast, prostate, etc.)

  * Note: Dural based metastases (e.g. commonly seen in breast cancer) are eligible
* Size of brain metastases

  * At least one intact metastasis (not previously treated with radiosurgery) must measure >= 2.0 cm and =< 4.0 cm in maximal extent on the contrasted pre-treatment magnetic resonance imaging (MRI) brain scan obtained =< 28 days prior to registration
  * If the largest lesion measures >= 2.0 to =< 4.0 cm in maximal extent the patient will be randomized
* Able to undergo contrast enhanced MRI brain
* Negative urine or serum pregnancy test completed =< 7 days prior to registration, for women of childbearing potential only
* Patient is willing and able to provide written informed consent or have a legally Authorized Representative (LAR) who is responsible for the care and well-being of the potential study participant provide consent.
* Karnofsky performance status (KPS) >= 50
* Eastern Cooperative Oncology Group (ECOG) performance score of (PS) >= 2
* Past radiosurgery or resection is allowed as long as no definitive evidence of progression in these locations

  * Note: Repeat radiosurgery to the same location/lesion is not allowed on this protocol

Exclusion Criteria:

* Any patient who has received previous whole brain radiation
* Any brain metastasis that is located in the brainstem measuring >= 2.0 cm in maximal extent
* Any patient with definitive evidence of leptomeningeal metastasis (LMD)

  * NOTE: For the purposes of exclusion, LMD is a clinical diagnosis, defined as positive cerebrospinal fluid (CSF) cytology and/or unequivocal radiologic or clinical evidence of leptomeningeal involvement. Patients with leptomeningeal symptoms in the setting of leptomeningeal enhancement by imaging (MRI) would be considered to have LMD even in the absence of positive CSF cytology, unless a parenchymal lesion can adequately explain the neurologic symptoms and/or signs. In contrast, an asymptomatic or minimally symptomatic patient with mild or nonspecific leptomeningeal enhancement (MRI) would not be considered to have LMD. In that patient, CSF sampling is not required to formally exclude LMD, but can be performed at the investigator's discretion based on level of clinical suspicion
* Any patient with an intact brain metastasis measuring > 4.0 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Time to local failure or symptomatic radiation brain necrosis of large brain metastasis | Up to 5 years
  Will determine if the composite endpoint of time to local failure or symptomatic radiation brain necrosis of a large brain metastasis [cumulative treatment failure (CTF)] is increased with fractionated stereotactic radiosurgery (FSRS) compared to single fraction stereotactic radiosurgery (SSRS).

SECONDARY OUTCOMES:
Overall survival (OS) | From study entry to death from any cause, assessed up to 5 years
  OS will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms. Medians and 95% confidence intervals will be reported.
Incidence of adverse events | Up to 2 years post radiation therapy
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.
Rates of radiation necrosis | Up to 5 years
  Will compare rates of radiation necrosis in patients who receive FSRS to patients who receive SSRS. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.
Central nervous system (CNS) failure patterns (Fractionation) | Up to 5 years
  Will evaluate if there is any difference in CNS failure patterns (e.g. local, distant brain failure) in patients who receive FSRS compared to patients who receive SSRS. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.
Time to neurologic death | Up to 5 years
  Will ascertain whether FSRS prolongs time to neurologic death as compared to SSRS. This will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms. Medians and 95% confidence intervals will be reported.
Quality of life (QOL) | Up to 5 years
  Will determine whether there are improved patient reported outcomes (Functional Assessment of Cancer Therapy [FACT]-Brain Symptom Index [FBrSI]-24) including quality of life for patients who receive FSRS compared to patients who receive SSRS. Changes over time in QOL from baseline will be compared between arms using the 2-sample t-test (or Wilcoxon Rank-Sum test for non-normal data). Box-plots will be used to show differences between arms graphically.
CNS failure patterns (Gamma Knife) | Up to 5 years
  Will evaluate if there is any difference in CNS failure patterns (e.g. local, distant brain failure) and symptomatic radiation necrosis rates in patients who are treated with Gamma Knife compared to patients who are treated with a linear accelerator platform. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.
Per lesion analysis between treatment arms: time to local failure | Up to 5 years
  Will determine whether differences in time to local failure differs between treatment arms (or other patient or treatment factors) when analyzed on a "per lesion" basis rather than the per patient basis utilized for the primary endpoint. Time-to-event models (Cox and Kaplan- Meier) with sandwich estimators for covariance will be utilized to in treatment comparisons, with model comparisons completed through log-likelihood and Akaike Information Criterion.
Per lesion analysis between treatment arms: time to necrosis | Up to 5 years
  Will determine whether differences in time to necrosis differs between treatment arms (or other patient or treatment factors) when analyzed on a "per lesion" basis rather than the per patient basis utilized for the primary endpoint. Time-to-event models (Cox and Kaplan- Meier) with sandwich estimators for covariance will be utilized to in treatment comparisons, with model comparisons completed through log-likelihood and Akaike Information Criterion.
Per lesion analysis between treatment arms: endpoint CTF | Up to 5 years
  Will determine whether differences in the composite endpoint CTF differs between treatment arms (or other patient or treatment factors) when analyzed on a "per lesion" basis rather than the per patient basis utilized for the primary endpoint. Time-to-event models (Cox and Kaplan- Meier) with sandwich estimators for covariance will be utilized to in treatment comparisons, with model comparisons completed through log-likelihood and Akaike Information Criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Brown, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials